CLINICAL TRIAL: NCT05506618
Title: A Multicenter COVID-19 Study Conducted to Evaluate the Performance of the LumiraDx SARS-CoV-2 Ag ULTRA Test at Point of Care Testing Sites
Brief Title: Performance Evaluation of LumiraDx COVID-19 (SARS-CoV-2) Ag ULTRA Test (ASPIRE-2)
Acronym: ASPIRE-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00053
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Subject are asked to provide nasal swab or nasopharyngeal swab samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Group A: Sample Collection (Other): 2x Nasopharyngeal Swab Sample Collection
  Interventions: Diagnostic Test: Nasopharyngeal swab
- Group B: Sample Collection (Other): 1x Nasopharyngeal Swab and 2x Nasal Swab Sample Collection
  Interventions: Diagnostic Test: Nasal Swab; Diagnostic Test: Nasopharyngeal swab
- Group C: Sample Collection (Other): 1x Nasopharyngeal Swab and 2x Nasal Swab Sample Collection for sample pooling
  Interventions: Diagnostic Test: Nasal Swab; Diagnostic Test: Nasopharyngeal swab
- Group D: Sample Collection (Other): 2x Nasal Swab Sample Collection
  Interventions: Diagnostic Test: Nasal Swab

INTERVENTIONS:
Diagnostic Test: Nasal Swab — Collection of one more nasal swabs
  Arms: Group B: Sample Collection; Group C: Sample Collection; Group D: Sample Collection
Diagnostic Test: Nasopharyngeal swab — Collection of one more nasopharyngeal swabs
  Arms: Group A: Sample Collection; Group B: Sample Collection; Group C: Sample Collection

SUMMARY:
Performance of the LumiraDx SARS-CoV-2 Ag ULTRA assay will be assessed by comparison to a reference method

DETAILED DESCRIPTION:
The study is a prospective, multi-center study. One (1) reference laboratory and approximately six (6) geographically diverse POC (Point of Care) locations (e.g. physician office laboratories, urgent cares, emergency departments, outpatient clinics, drive through testing sites or research centers) in the U.S. will participate in the study. Testing in the reference laboratory will be performed by trained laboratory personnel. Testing at the POC sites will be performed by non-laboratory health professionals who are representative of typical intended use operators (e.g. nurses, physician assistants, medical assistants, etc.). Each site will have a minimum of one (1) untrained intended use operator who will perform testing under this protocol.

A subject's participation in this study will consist of a single visit. Following completion of the informed consent process and a review of Inclusion/Exclusion criteria to determine eligibility, each subject will receive a unique study identification number.

Subjects will have nasopharyngeal or nasal or throat swabs collected. Specimens will be obtained from each subject enrolled using standard collection methods.

The LumiraDx SARS-CoV-2 Ag ULTRA Test will be performed at POC sites by intended use operators (e.g. nurses, physician assistants, medical assistants, etc.). Each site will have a minimum of one (1) untrained intended use operator who will perform testing under this protocol.

The LumiraDx SARS-CoV-2 Ag ULTRA Test will be performed at the site on the same day as the date of collection using one swab for each subject enrolled. A central laboratory will perform reference testing.

Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) will be estimated for the LumiraDx SARS-CoV-2 Ag ULTRA Test results as compared with the reference Test.

A minimum of thirty (30) positive SARS-CoV-2 are required, but it is likely because of the prevalence of SARS-CoV-2 in the population, that a greater number of negatives will be obtained during the prospective collection of positive samples; therefore, approximately four-hundred (400) subjects will be enrolled. A minimum of thirty (30) negative samples are required.

ELIGIBILITY:
Inclusion Criteria

1. Subject may be of any age or gender.
2. Preliminary assessment of the subject by the Investigator/designee should be suggestive of COVID-19 at the time of the study visit. The subject must present as symptomatic, meaning they have exhibited one or more of the following signs and symptoms for eligibility: fever, cough, shortness of breath, difficulty breathing, muscle pain, headache, sore throat, chills, repeated shaking with chills, new loss of taste or smell congestion or runny nose, diarrhea, nausea or vomiting. The onset of these symptoms will be recorded and will be within the last twelve (12) days.

   or The subject is asymptomatic and is neither currently exhibiting signs or symptoms of SARS-CoV-2 nor has experienced signs or symptoms within the past fourteen (14) days, and has not knowingly been exposed to someone with a positive test result within the last fourteen (14) days
3. Participant (or parent/legal guardian) capable and willing to give informed consent/assent.

Exclusion Criteria

1. The subject underwent a nasal wash/aspirate as part of standard of care testing during this study visit.
2. The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
3. Subjects undergoing treatment currently and/or within the past thirty (30) days of the study with medication to treat novel Coronavirus SARS-CoV-2 like illness symptoms, which may include but is not limited to Remdesivir or convalescent plasma therapy for SARS-CoV-2.
4. The subject has previously participated in this research study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Performance Evaluation | 4 months
  Evaluation of performance of the device versus a reference method using standard qualitative comparison techniques (Percent Agreement)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Girgis, MD, Principal Investigator — Advanced Investigative Medicine; Michael Vaughn, MD, Principal Investigator — Cahaba Research, Inc.; Frank Calcagno, MD, Principal Investigator — Cyn3rgy Research; Hilda Brito, MD, Principal Investigator — Healthy Life Research, Inc.; Rogelio Machuca, MD, Principal Investigator — The Machuca Foundation, Inc.; Tewodros Teketel, MD, Principal Investigator — Zion Urgent Care
Locations (6):
- United States (6):
  - Cahaba Research, Inc., Birmingham, Alabama
  - Advanced Investigative Medicine, Hawthorne, California
  - Healthy Life Research, Inc., Miami, Florida
  - The Machuca Foundation, Inc., Las Vegas, Nevada
  - Cyn3rgy Research, Gresham, Oregon
  - Zion Urgent Care, Katy, Texas

IPD SHARING:
Plan to Share IPD: No